CLINICAL TRIAL: NCT04544800
Title: Development of Upper Aerodigestive Tract Splint
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Relocation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-5577
Record Dates: First submitted 2020-08-26; First posted 2020-09-10 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Splints
Keywords: Upper Aerodigestive Tract; Visualization; Surgical Instrumentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of Splint for UADT Visualization (Experimental): Use of device to view UADT
  Interventions: Device: Use of Splint for UADT Visualization

INTERVENTIONS:
Device: Use of Splint for UADT Visualization — The use of a splint to assist the patient and the surgeon with UADT procedures.

SUMMARY:
The study hypothesis is that a splint will improve access to the upper aerodigestive tract (UADT) for diagnosis and treatment.

DETAILED DESCRIPTION:
This is a pilot study of 30 patients. We will tabulate the data for efficacy, there will be no statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Require a procedure involving the upper aerodigestive tract (UADT)

Exclusion Criteria:

* Prior surgery to tongue or mouth that precludes the use of the splint
* Trismus with mouth opening that does not allow for use of the splint
* TMJ dysfunction that precludes the use of the splint
* Allergy to local anesthetic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Patient Splint Satisfaction Questionnaire | Immediately after the intervention/procedure/surgery
  Self-administered, 6-item questionnaire to evaluate splint satisfaction.
Physician Splint Satisfaction Questionnaire | Immediately after the intervention/procedure/surgery
  A 14-item questionnaire to evaluate the surgeon satisfaction with the splint.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas B Chepeha, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada